CLINICAL TRIAL: NCT05208099
Title: Study of the Immunomodulation of the Immune Response in Hidradenitis Suppurativa and in Vitro and ex Vivo Evaluation of a New Therapeutic Strategy (IMOHS)
Brief Title: Study of the Immunomodulation in the Hidradenitis Suppurativa and Evaluation of a New Therapeutic Strategy
Acronym: IMOHS
Status: Not yet recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P00111
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; inflammatory nodules; abscesses; fistulas; scars; surgery
MeSH Terms: conditions — Hidradenitis Suppurativa; Abscess; Fistula; Cicatrix | interventions — Hematologic Tests; Abdominoplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Hidradenitis suppurativa
  Interventions: Biological: Blood tests; Procedure: exeresis
- Controls (coming for abdominoplasty)
  Interventions: Procedure: abdominoplasty

INTERVENTIONS:
Biological: Blood tests — For patients, it will be performed:
  * a collection of blood samples (3 tubes of 5 mL) according to the usual medical management, in order to search for cardiovascular comorbidities associated with HS,
  * A collection of 3 EDTA tubes and 2 additional dry tubes of 5 mL each according to the needs of the study.
  Groups: Patients with Hidradenitis suppurativa
Procedure: exeresis — For patients, it will be performed:
  - 6 tissue samples from the total excision specimen: two samples from the acute inflammatory zone (nodule, abscess, fistula) of 1 cm3; two samples from the chronic lesion zone (scar) of 1 cm3 and two samples from the peri-lesion zone (in the margin) of 1 cm3 on fresh tissue.
  Groups: Patients with Hidradenitis suppurativa
Procedure: abdominoplasty — For the controls, 6 fresh skin samples of 1 cm3 each will be taken from the abdominoplasty operation:
  * four in the center,
  * two in the margin
  Groups: Controls (coming for abdominoplasty)

SUMMARY:
Hidradenitis suppurativa (HS), also known as Verneuil's disease, is a chronic inflammatory dermatosis of the hair follicule located mainly in the skin folds (axillae, inguinal, submammary, etc.).

Currently, treatments are mainly limited to the use of broad-spectrum antibiotics in order to control outbreaks of hidradenitis suppurativa. Surgical treatment is the only curative treatment, but requires disfiguring removals with major scarring consequences.

Pathophysiologically, HS appears to be a primary abnormality of the pilosebaceous-apocrine unit, causing follicular occlusion, followed by the development of perifollicular cysts with commensal bacterial overgrowth, and finally rupture into the dermis causing an exaggerated inflammatory response. At present, few studies have examined the role of the regulatory immune system and its involvement in this disease.

We are also interested in analyzing the impact of new therapeutic strategies on hidradenitis suppurativa, and more particularly the impact of photodynamic therapy (PDT) which is a technique that has been used for a long time in dermatology, notably for the treatment of precancerous and cancerous lesions.

This technique has shown interesting results on inflammatory dermatoses such as acne.

This research consists in studying the immunomodulation of the immune response in HS and in evaluating a new therapeutic strategy based on PDT alone or in combination with antimicrobial peptides (PAMs).

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS), also known as Verneuil's disease, is a chronic inflammatory dermatosis of the hair follicule located mainly in the skin folds (axillae, inguinal, submammary, etc.). The disease is characterized by pain, inflammatory nodules, abscesses, fistulas and hypertrophic " rope " scars that considerably alter the quality of life of patients.

Currently, the treatment is mainly limited to the use of broad-spectrum antibiotics in order to control the outbreaks of HS. This medical treatment is currently controversial because of the risk of inducing bacterial resistance. Surgical treatment is the only curative treatment, but requires disfiguring removals with major scarring consequences.

Pathophysiologically, HS appears to be a primary abnormality of the pilosebaceous-apocrine unit, which causes follicular occlusion, followed by the development of perifollicular cysts with commensal bacterial proliferation, and finally rupture into the dermis causing an exaggerated inflammatory response. At present, few studies have examined the role of the regulatory immune system and its involvement in this disease.

In the context of HS, it has recently been shown from patient samples that there is an abnormality concerning the stem cells present in the follicular bulb. It can be asked whether the abnormalities observed in hair follicle stem cells of HS patients could be the source of pro-inflammatory exosomes playing a role in HS flares.

The impact of new therapeutic strategies on hidradenitis suppurativa, and more particularly the impact of photodynamic therapy (PDT) which is a technique used for a long time in dermatology, notably for the treatment of precancerous and cancerous lesions will be also evaluated.

This technique has shown interesting results on inflammatory dermatoses such as acne with an " antibiotic " effect.

Thus, this research consists in studying the immunomodulation of the immune response in HS and in evaluating a new therapeutic strategy based on PDT alone or in combination with antimicrobial peptides (PAMs). This is a prospective observational multicenter study of type 3. This study is composed of two steps : first an in vitro part, secondly an ex vivo part allowing to validate the results obtained in vitro on human samples.

ELIGIBILITY:
Inclusion criteria for HS patients :

* Adult patients (≥18 years)
* Carrier of moderate to severe (Hurley grade ≥2) hidradenitis suppurativa of classical or gluteal phenotype
* Having an indication for surgical treatment (indication for excision)
* Not receiving immunomodulatory treatments (corticotherapy, biotherapy, apremilast, retinoids) or immunosuppressive treatments (methotrexate, ciclosporin) in the 6 months before inclusion, excluding antibiotics
* Agreement to participate
* Affiliated to social security

Inclusion criteria for control receiving abdominoplasty :

* Adult patients (≥18 years)
* With no history of hidradenitis suppurativa or lesions suggestive of hidradenitis suppurativa (recurrent fold abscesses, recurrent fold suppuration, repeated draining in fold areas)
* With an indication for abdominoplasty surgery
* Not receiving immunomodulatory treatments (corticotherapy, biotherapy, apremilast, retinoids) or immunosuppressive treatments (methotrexate, ciclosporin) in the 6 months preceding inclusion, excluding antibiotics
* Agreement to participate
* Affiliated to social security

Criteria for non-inclusion of patients with HS :

* Immunosuppression, autoimmune disease(s), cancerous disease, or acute or chronic infectious disease
* Difficulty understanding or reading French
* Patients already included in a therapeutic interventional trial
* Patients under guardianship or curatorship
* Pregnant or breast feeding women
* Syndromic hidradenitis suppurativa, hidradenitis suppurativa of follicular phenotype

Criteria for non-inclusion of controls receiving abdominoplasty :

* Immunosuppression, autoimmune disease(s), cancerous disease, or acute or chronic infectious disease
* Difficulty understanding or reading french
* Patients already included in a therapeutic interventional trial
* Patients under guardianship or curatorship
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with hidradenitis suppurativa and subjects without hidradenitis suppurativa undergoing abdominoplasty
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of different types of immune cell populations | Day 0
  Prevalence of cell populations will be determined by cytometry
Activation of lymphocytes | Day 0
  The activation state of circulating lymphocytes will be analyzed by flow cytometry using antibodies coupled to fluorochromes specifically targeting the following membrane markers: CD4, CD30, CD69, Anti-HLADR, CD152, CD197, CD25, CD8.
Prevalence of innate lymphoid cells | Day 0
  The prevalence of innate lymphoid cells will be determines by cytometry
Gene expression analysis | Day 0
  A microarray assay will be performed in order to determine the expression of genes of interest.
Secretome analysis | Day 0
  The pg/mL concentrations of different cytokines in the serum of HS patients versus healthy controls will be determined using ELISA (Luminex™) in order to be able to determine the differences in activation of immune pathways : Th1/Th2, Th9/Th17/Th22/Treg, inflammatory cytokines, Immunosuppressive cytokine.

SECONDARY OUTCOMES:
Size of exosomes | Day 0
  The size of exosomes will be measured by the Tunable resistive Pulse sensing method
Concentration of exosomes | Day 0
  The concentration of exosomes will be measured by the Tunable resistive Pulse sensing method
Quantification of antimicrobial peptides | Day 0
  Several antimicrobial peptides such as elafin/SHALP, dermcidin, S100A7/psoriasin, S100A8/calgranulin A, S100A9/calgranulin B, LL-37 (cathelicidin), h-βd1, h-βd2, h-βd3, h-βd4, ribonuclease 7, SLPI/ALP from HS patient serum versus blood baqs (control) as well as in supernatants of HS lesion tissue versus abdominoplasty tissue (control) cultured in microslices will be quantified by ELISA
Quantification of wound healing | Day 0
  Wound healing capacity
  We will evaluate the ability to restore wound healing in in vitro HS models (HaCaT NCSTN-/-line) versus the healthy model (HaCaT wild type) by performing wound healing and migration assays (IBIDI) with and without the addition of exogenous PAMs lacking in HS.
Efficacity of the Photodynamic Therapy (PDT) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Marie LAMIAUX, Principal Investigator — Lille Catholic University
Locations (2):
- France (2):
  - Hôpital Saint Vincent-de-Paul, Service de Dermatologie-Vénéréologie, Lille
  - Hôpital Saint Philibert - Service de Chirurgie Viscérale, Lomme

IPD SHARING:
Plan to Share IPD: No